CLINICAL TRIAL: NCT05063461
Title: Evaluation of the Analgesia Nociception Index With Varying Remifentanil Concentrations Under Sevoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Changwei Wei, Deputy chief physician, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00375930
Record Dates: First submitted 2021-09-15; First posted 2021-10-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sevoflurane with different site effect concentrations of remifentanil (Experimental): The tetanic stimulus is conducted between laryngeal mask intubation and surgical stimulation, while no other noxious stimuli are presented. The effect site concentration of remifentanil is increased step-by-step via a Target Controlled infusion device to a concentration of 2, 4, 6 ng/ml. At least 5min of the steady-state period is maintained before tetanic stimulus.
  Interventions: Device: Tetanic stimulation; Procedure: Skin incision

INTERVENTIONS:
Device: Tetanic stimulation — For each participant, record the first concentration that ANI≥50 after the tetanic stimuli, as the sufficient concentration.
Procedure: Skin incision — Infuse the sufficient concentration for at least 5min of the steady-state period, then surgical stimulus is applied. The surgical stimulus is defined as the first skin incision to establish pneumoperitoneum.

SUMMARY:
Analgesia Nociception Index（ANI）which is derived from heart rate variability can be used to detect noxious stimulation during propofol while changing remifentanil concentrations. The aim of this study is to verify the effectiveness of ANI predictability for actual surgical noxious stimuli while satisfying the individual analgesic status by pre-tetanus-induced ANI determination during sevoflurane while changing remifentanil concentrations.

DETAILED DESCRIPTION:
General anesthesia with sevoflurane and remifentanil is widely used in minor surgeries. Monitoring noxious stimulation during general anesthesia is still worth further studies and reaching clinical consensus. Analgesia Nociception Index can be used to detect noxious stimulation during propofol while changing remifentanil concentrations. Previous studies suggest that an ANI≥50 can be useful in detecting sufficient analgesia for patients who cannot self-report pain. The aim of this study is to verify the effectiveness of ANI predictability for actual surgical noxious stimuli while satisfying the individual analgesic status by pre-tetanus-induced ANI determination during sevoflurane while changing remifentanil concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18- 65 years
* ASA physical status I or II
* Elective surgery in general anesthesia planned
* Written informed consent

Exclusion Criteria:

* Use of CNS-active medication or abuse of alcohol
* Presents of any neuromuscular or neurologic disease
* History of cardiac arrhythmia
* Pregnancy or using a pacemaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
To verify the effectiveness of ANI predictability for actual surgical noxious stimuli while satisfying the individual analgesic status by pre-tetanus-induced ANI determination. | Change from Baseline ANI that 2 minutes after applied tetanic stilumation
  Tetanic stimulations are applied at different effect site concentrations of remifentanil under sevoflurane anesthesia. ANI is range from 0-100. Bigger number means better analgesic level. ANI≥50 is considered to be under adequate analgesia. Tetanic stimulation is a standard tester of nociceptive stimulus. The number of ANI will fall down if the patient is feeling pain.

SECONDARY OUTCOMES:
The ANI predictability for tetanic noxious stimuli | Change from Baseline Systolic Blood Pressure that 2 minutes after applied tetanic stilumation
  ANI is range from 0-100. Bigger number means better analgesic level. ANI≥50 is considered to be under adequate analgesia. The number of ANI will fall down if the patient is feeling pain.
The heart rate predictability for tetanic noxious stimuli | Change from Baseline Heart Rate that 2 minutes after applied tetanic stilumation
  Heart Rate will go up if patient is feeling pain.
The Bispectral Index predictability for tetanic noxious stimuli | Change from Baseline Bispectral Index that 2 minutes after applied tetanic stilumation
  Bispectral Index will go up if patient is feeling pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yang L, Wang X, Wen H. Evaluation of the effectiveness of analgesia nociception index (ANI) predictability for surgical stimuli under personal analgesic sufficiency status (PASS) measured by pre-tetanus-induced ANI: a pilot study. J Clin Monit Comput. 2023 Dec;37(6):1585-1591. doi: 10.1007/s10877-023-01044-y. Epub 2023 Jul 7. PMID 37418059